CLINICAL TRIAL: NCT02322359
Title: Impact of a Feedback Device, CPRmeter®, on Chest Compression Quality During Extend Cardio-pulmonary Resuscitation. A Manikin Study.
Brief Title: Compression Is Life In Cardiac Arrest - Fatigue Study
Acronym: CILICA-FS
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: A14-D20-VOL.21
Record Dates: First submitted 2014-11-27; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Context: Chest compressions represent an important physical effort leading to fatigue and cardiopulmonary resuscitation quality degradation. Despite a known harmful effect of chest compressions interruptions, current guidelines still recommend provider switch every 2 minutes. Feedback impact on chest compressions quality during an extended cardiopulmonary resuscitation remains to be assessed.

Study design: simulated prospective monocentric randomized crossover trial. Participants and methods: Sixty professionals rescuers of the pre-hospital care unit of University Hospital of Caen (doctors, nurses and ambulance drivers) are enrolled to performed 10 minutes of continuous chest compression on manikin (ResusciAnne®, Laerdal), twice, with and without a feedback device (CPRmeter®). Correct compression score (the main criterion) is defined by reached target of rate, depth and leaning at the same time (recorded continuously).

Hypothesis: Feedback device delay fatigue effect arises during cardiopulmonary resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Operational staff of University hospital of Caen pre-hospital unit

Exclusion Criteria:

* medical contraindication
* refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers from University hospital of Caen pre-hospital unit
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Correct compression score | 24h
  Correct compression score is defined by reached target of rate, depth and leaning at the same time

SECONDARY OUTCOMES:
Decrease time of 30% of correct compression score | 24h
chest compression deep | 24h
chest compression rate | 24h
percentage of chest compression without leaning | 24h
percentage of chest compression with correct deep | 24h
percentage of correct chest compression rate | 24h
participants' fatigue (Borg's scale) | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Clement BULEON, MD, Principal Investigator — University Hospital of Caen
Locations (1):
- University Hospital of Caen, Caen, France